CLINICAL TRIAL: NCT01705652
Title: Phase II Study to Assess the Activity of Nexrutine® in Prostate Cancer Patients Undergoing Surgery or Radiation Therapy
Brief Title: Study to Assess the Activity of Nexrutine® in Prostate Cancer Patients
Acronym: Nexrutine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of funding
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Gregory P. Swanson, MD, Clinical Professor, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20100308H
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
Keywords: nexrutine; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nexrutine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nexrutine Surgery Group (Experimental): Surgery Group: Nexrutine 500mg by mouth, three times per day, given prior to surgery.
  Interventions: Drug: Nexrutine
- Nexrutine Radiation Group (Experimental): Radiation Group: Nexrutine 500mg by mouth, three times per day, given prior to and during radiation treatment.
  Interventions: Drug: Nexrutine

INTERVENTIONS:
Drug: Nexrutine — Nexrutine 500mg by mouth, three times per day, given prior to surgery or prior to and during radiation treatment.
  Other Names: bark extract of Phellodendron amurense

SUMMARY:
The purpose of the study is to (1) to determine the rate of PSA decline (the number declining). Tissue will be obtained for ancillary studies and (2) to determine the number of patients with a PSA decline to <1.0 ng/ml at 3 months in patients receiving Nexrutine® with standard radiation therapy. The Secondary Objective is to confirm the tolerability of this regimen. The Third Objective (Ancillary studies) is To evaluate the molecular response of Nexrutine®. Molecular response is defined as changes in the molecular pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologic diagnosis of prostate cancer (in more than 1 core) with one of the following:

   * Gleason > 6,
   * Unilateral Gleason 6 in ≥ 3 cores,
   * bilateral Gleason 6,
   * PSA > 10.0 ng/ml.
2. Age ≥18 years.
3. Has an ECOG Performance Status 0-2 or Karnofsky 60-100.
4. Has the following laboratory values at study entry: absolute neutrophil count (ANC) ≥ 1,500 cells/μL; platelet count ≥ 100,000 cells/μL; hemoglobin ≥ 9 g/dL; total serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); ALT and AST ≤ 1.5 x institutional ULN if alkaline phosphatase is ≤ULN creatinine and BUN ≤ 1.5 x institutional upper limit of normal (ULN)
5. Signed informed consent
6. No new, undiagnosed bone pain or has a negative bone scan. (within 2 months of consent) If there is no bone pain, then a bone scan is not required.

Exclusion Criteria:

1. Has documented metastatic disease.
2. Has received a prior chemotherapy or androgen ablation.
3. Has received prior immunotherapy.
4. Has been previously treated with Strontium, Samarium, other systemic radioisotopes or radiation therapy.
5. Has diagnosis of congestive heart failure
6. Currently taking anticoagulation medications, i.e., coumadin or heparin. Over the counter aspirin and ibuprofen are allowed.
7. Is receiving any other investigational agents for cancer.
8. Has a history of other malignancy within the last 5 years, which could affect the diagnosis or assessment of prostate cancer.
9. Has a serious intercurrent illness with a life expectancy of less than 5 years.
10. Has a concomitant medical, psychological, or social circumstance, which would interfere with compliance with the protocol treatment and follow-up.
11. Use of any herbal or alternative regimens, which may have antineoplastic or hormonal activity (including but not limited to finasteride, dutasteride, Saw Palmetto, PC-SPES, shark cartilage, etc), is prohibited while receiving study treatment.
12. Clinical stage T3 or T4 and PSA >10 ng/ml and Gleason > 8.
13. Patient is to receive adjuvant androgen ablation with the radiation.
14. EKG which shows a baseline QTc > 450 msec or ischemic changes. For ischemic changes, patient will be eligible if evaluated and cleared by internal medicine.
15. Previous history of drug-induced QTc prolongation and/or concurrent treatment with medications that are known to produce or are suspected of QT prolongation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Swanson, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; William E. Jones, III, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio and ALM VA Hospital
Locations (1):
- The University of Texas Health Science Center at San Antonio, study site: ALM VA Hospital, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 7/20/2011 to 4/16/2013 from the ALM VA South Texas urology clinic.
Pre-assignment Details: Subjects were required to have a diagnosis of prostate cancer and treatment planned by surgery or radiation therapy.. Subjects were excluded if they were currently taking anticoagulation medications, or medications that are known to produce or are suspected of QT prolongation.
Period: Overall Study
Arm/Group | Nexrutine Surgery Group | Nexrutine Radiation Group
Started | 9 | 12
Completed | 6 | 9
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — non-compliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nexrutine Surgery Group: Surgery Group: Nexrutine 500mg by mouth, three times per day, given prior to surgery. Minimum of 30 days and maximum of 80 days before surgery. The final dose is taken the day before surgery.
- Nexrutine Radiation Group: Radiation Group: Nexrutine 500mg by mouth, three times per day, given prior to and during radiation treatment. Minimum of 30 days and maximum of 60 days prior to the start of radiation therapy and then during treatment. The final dose is taken the last day of radiation.
- Total: Total of all reporting groups
Arm/Group | Nexrutine Surgery Group | Nexrutine Radiation Group | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: PSA (Prostate Specific Antigen)
Description: PSA decline to < 1.0 ng/ml at 3 months post end of radiation or surgery
Time Frame: 3 months post end of radiation treatment or surgery
Population: Radiation Group: One subject who did not complete the study was included as he did stay in the study through the 3 month post radiation treatment time period, and dropped out after that time.
Measure: Number; unit: participants
Groups:
- Radiation Group: Nexrutine by mouth three times per day for a minimum of 30 days and a maximum of 60 days prior to the start of radiation therapy and during treatment. The final dose will be taken the last day of radiation.
- Surgery Group: Nexrutine by mouth three times per day prior to surgery for a minimum of 30 days and maximum of 80 days. The final dose is taken the day before surgery.
Arm/Group | Radiation Group | Surgery Group
Number analyzed (Participants) | 10 | 6
participants | 2 | 6

ADVERSE EVENTS:
Time Frame: During Treatment plus 30 days.
Description: Regular investigator assessment, regular laboratory testing
Arm/Group | Nexrutine Surgery Group | Nexrutine Radiation Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 9/9 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nexrutine Surgery Group (N=9) | Nexrutine Radiation Group (N=12)
Anemia (Blood and lymphatic system disorders) | 7 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Burn (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 9
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
EKG QT corrected interval prolongation (Investigations) | 1 | 2
Edema limbs (General disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 1 | 6
Flatulence (Gastrointestinal disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4
Hypotension (Vascular disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1
Platelet count decreased (Investigations) | 2 | 3
Proctitis (Gastrointestinal disorders) | 0 | 5
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Urine discoloration (Renal and urinary disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Weight gain (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspatrate aminotransferase increased (Investigations) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 2 | 0
Creatinine increased (Investigations) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No